CLINICAL TRIAL: NCT06698653
Title: Assessment of the Benefit of the Mobility Assistance System (SAM) on Transfer Independence for a Reimbursement Request
Acronym: SAM-24
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WINNCARE (Industry)
Collaborators: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-A01608-39
Record Dates: First submitted 2024-11-18; First posted 2024-11-21 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: no Specific Condition Targeted

STUDY DESIGN:
Intervention Model Description: Group 1 (phase A = experimental (7 days), then phase B= control (7 days)) Group 2 (phase B = control (7 days), then phase A = experimental (7 days))
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase A : Experimental (Experimental): Phase A corresponds to the experimental phase where the patient will use the experimental device during 7 days.
  Interventions: Device: SAM device (experimental): a removable structure, fixed to the horizontal frame of the medical bed, equipped with a handle to assist the sitting-up process
- Phase B : Control (Active Comparator): Phase B corresponds to the control phase where the patient will use the control device during 7 days.
  Interventions: Device: Over bed pole hoist (control device)

INTERVENTIONS:
Device: SAM device (experimental): a removable structure, fixed to the horizontal frame of the medical bed, equipped with a handle to assist the sitting-up process — The patients will use the experimental device during 7 days straight as well as the comparator during 7 days straight. The order in which they will use each device will depend on the groupe they have been randomized in : - Groupe 1 : Experimental device during 7 days then control device during 7 days - Groupe 2 : Control device during 7 days then experimental device during 7 days
  Arms: Phase A : Experimental
Device: Over bed pole hoist (control device) — The patients will use the experimental device during 7 days straight as well as the comparator during 7 days straight. The order in which they will use each device will depend on the groupe they have been randomized in : - Groupe 1 : Experimental device during 7 days then control device during 7 days - Groupe 2 : Control device during 7 days then experimental device during 7 days
  Arms: Phase B : Control

SUMMARY:
This is a randomized, cross-over, multi-center, intention-to-treat, open-label study to assess the impact of the SAM Ergonom light (SAM) device on independence when transferring from the supine to the sitting position at the edge of the bed in a population of individuals with an inability to transfer independently from the supine to the sitting position in bed, compared with the use of a raising arm.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Unable to transfer from lying to sitting independently
* Requiring technical assistance or the help or supervision of a third party
* Using a medical bed
* In-patient care for a minimum of 3 weeks in a medical or rehabilitation facility
* Having freely consented to participate
* Affiliated with a social security scheme or entitled to benefits

Exclusion Criteria:

* Non-consolidated spinal or pelvic fracture
* Degenerative shoulder
* Cardiovascular disorders caused by physical exertion
* Joint pain localized to dorsolumbar spine
* Behavioural disorders (opposition, agitation, dementia)
* Invalid patient (disability, low tonicity), agitated, not lucid (confused, disoriented) at risk of falling, requiring physical restraint with bed rails on medical prescription
* Functional inability to move independently
* Cognitive impairment affecting reliability of response to questionnaires
* Motor or algic incapacity of the 2 upper limbs not allowing the use of a technical aid (lifting frame or SAM) to ensure transfer from lying to sitting position in bed
* Patient less than 146 cm tall
* Patient weighing less than 30 kg or more than 200 kg
* Patient with a mattress incompatible with the OS'CARE device
* Mattress length less than 190 cm or greater than 200 cm, and width less than 85 cm or greater than 120 cm

In addition, vulnerable persons covered by articles L. 1121-5 to 8 and L. 1122-1-2 of the French Public Health Code are excluded from the study:

* Pregnant, parturient or breast-feeding women
* Persons deprived of their liberty by judicial decision (including guardianship, curatorship and safeguard of justice) or administrative decision
* Persons under psychiatric care or admitted to a health or social institution for purposes other than research.
* Person in an emergency situation unable to give prior consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The impact on transfer independence will be measured by comparing the "bed transfer" item of the Functional Independence Measure (FIM), carried out at D7 and D14 by direct observation of the participant by the therapist. | At day 7 and day 14 of the experiment

SECONDARY OUTCOMES:
The psychosocial impact, including quality of life, will be measured by comparing the scale for measuring the psychosocial impact of a technical aid (F-PIADS) at D7 and D14. | At day 7 and day 14 of the experiment
Satisfaction with the use of the SAM device will be measured by comparing the satisfaction scale with the technical aid (ESAT) at D7 or D14. | At day 7 and day 14 of the experiment
Device acceptability will be measured by a questionnaire based on the Unified Theory of Acceptance and Use of Technology (UTAUT) model at D7 and D14. | At day 7 and day 14 of the experiment
Overall independence will be measured by comparing global FIM at D7 and D14. | At day 7 and day 14 of the experiment
Effort during supine-to-sitting transfers will be measured by comparing the duration of a supine-to-sitting transfer at the edge of the bed at D7 and D14, and by the average duration of the transfer during the period of use of the devices. | At day 7 and day 14 of the experiment
The quantity and quality of the transfer will be evaluated indirectly by the total number of lifts and attempted lifts from the bed over 7 days for each device, measured by OS'CARE bed presence sensors. | At day 7 and day 14 of the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Leblong, Principal Investigator — Fondation Saint Helier
Locations (3):
- France (3):
  - Centre Mutualiste de Rééducation et de Réadaptation Fonctionnelles (CMRRF) de Kerpape, Ploemeur
  - Fondation Ildys, Ploemeur
  - Pôle Saint Hélier, Rennes